CLINICAL TRIAL: NCT01146353
Title: Pharmacokinetic Assessment of Peramivir in Hospitalized Adults Undergoing Continuous Renal Replacement Therapy
Status: Withdrawn | Type: Observational
Why Stopped: Peramivir EUA terminated by FDA.
Sponsor: Midwestern University (Other)
Collaborators: Northwestern University (Other); BioCryst Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Marc Scheetz, Associate Professor, Midwestern University
Other Study IDs: STU00023343
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Influenza; Renal Failure
Keywords: peramivir; CVVH; CRRT; CVVHD; influenza; sieving coefficient; clearance
MeSH Terms: conditions — Influenza, Human; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRRT Patients receiving Peramivir: Eligible patients are male or female patients ≥18 years of age who are hospitalized, undergoing CVVH or CVVHD, and receiving peramivir.
  Eligible patients will additionally have the following: blood flow rate will be required to be ≥100 mL/ min with an ultrafiltrate +/- dialysis flow rate greater than or equal to 3000mL/hr, and the continuous renal replacement therapy must be scheduled to run for the full duration of the dosing interval (full 24 hours).
  Written informed consent in a form approved by the Northwestern University and the Midwestern University Institutional Review Boards will be granted by the patient.

SUMMARY:
Pharmacokinetics for peramivir have not been well characterized in patients undergoing continuous renal replacement therapy CRRT - either Continuous veno-venous hemofiltration (CVVH) +/- dialysis (CVVHD). CRRT is commonly utilized in the hospital setting for patients with acute kidney injury for metabolic correction, slow continuous fluid removal, and to maintain hemodynamic stability. CRRT commonly alters drug disposition and clearance, and dosing regimens often need alteration in patients receiving CRRT. Doses required to generate predictable serum concentrations can be calculated from known patient parameters such as replacement fluid and dialysate flow rate, sieving coefficients, and desired serum concentrations. However, pharmacokinetic studies must be performed in CRRT patients to generate drug removal constants or sieving coefficients. Of note, the clearance of drugs by conventional hemodialysis cannot be used to extrapolate clearances with CRRT secondary to differences in ultrafiltration rates and dialysis membranes. The investigators propose an open label study to obtain peramivir pharmacokinetics in patients undergoing CRRT.

DETAILED DESCRIPTION:
This study has been closed. No patients were enrolled as the peramivir EUA was rescinded.

ELIGIBILITY:
Inclusion Criteria

* Patient is hospitalized and undergoing continuous renal replacement therapy (CRRT) as a result of the clinical management of the patient (i.e. CRRT is not initiated for the purpose of this study).
* Patient is receiving peramivir for a positive rapid antigen test for influenza or on the basis of clinical suspicion with a high local epidemiological prevalence of H1N1 disease.
* Patient has a CRRT blood flow rate greater than or equal to 100 mL/min with an ultrafiltrate +/- dialysis flow rate greater than or equal to 3000mL/hr,
* The patient is anticipated to require CRRT and peramivir treatment for a full 24 hours (i.e. life expectancy is not less than 24 hours).

Exclusion Criteria

* The patient has received greater than 5 doses of peramivir.
* The subject has a pre-existing illness that, in the opinion of the investigator, would place the subject at an unreasonably increased risk through participation in this study.
* The patient is receiving CRRT utilizing a pre-membrane dilution method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are male or female patients ≥18 years of age who are hospitalized, undergoing CVVH or CVVHD, and receiving peramivir.
  Eligible patients will additionally have the following: blood flow rate will be required to be ≥100 mL/ min with an ultrafiltrate +/- dialysis flow rate greater than or equal to 3000mL/hr, and the continuous renal replacement therapy must be scheduled to run for the full duration of the dosing interval (full 24 hours).
  Written informed consent in a form approved by the Northwestern University and the Midwestern University Institutional Review Boards will be granted by the patient.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be to determine the sieving coefficient for peramivir. | upon study completion (estimated 2 yrs)

SECONDARY OUTCOMES:
Determine the extracorporeal clearance for peramivir | upon study completion (estimated 2 yrs)

CONTACTS AND LOCATIONS:
Overall Officials: Marc H Scheetz, PharmD, MSc, Principal Investigator — Midwestern University and Northwestern Memorial Hospital; Michael Ison, MD, Principal Investigator — Northwestern University
Locations (1):
- Midwestern University/Northwestern Memorial Hospital, Chicago, Illinois, United States